CLINICAL TRIAL: NCT02879578
Title: Safety and Tolerability Study of NBI-98854 for the Treatment of Subjects With Tourette Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-98854-1601
Record Dates: First submitted 2016-08-10; First posted 2016-08-25 (Estimated); Results first posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — valbenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Valbenazine (Children) (Experimental): Children (6 to 11 years of age) received valbenazine 10 mg once daily for 4 weeks. At the end of Week 4, investigators could escalate the dose to 20 mg or continue with the participant's current dose for the remainder of the treatment period.
  Interventions: Drug: Valbenazine
- Valbenazine (Adolescents) (Experimental): Adolescents (12 to 17 years of age) received valbenazine 20 mg once daily for 4 weeks. At the end of Week 4, investigators could escalate the dose to 40 mg or continue with the participant's current dose for the remainder of the treatment period.
  Interventions: Drug: Valbenazine
- Valbenazine (Adults) (Experimental): Adults (18 to 64 years of age) received valbenazine 40 mg once daily for 4 weeks. At the end of Week 4, investigators could escalate the dose to 80 mg or continue with the participant's current dose for the remainder of the treatment period.
  Interventions: Drug: Valbenazine

INTERVENTIONS:
Drug: Valbenazine
  Other Names: NBI-98854

SUMMARY:
Phase 2, open-label, fixed-dose titration study to evaluate the safety and tolerability of NBI-98854 administered once daily for a total of 24 weeks in children, adolescents, and adults with Tourette Syndrome (TS).

ELIGIBILITY:
Inclusion Criteria:

* Have participated in and completed the NBI-98854-1501 (T-Force Green) or NBI-98854-1505 (T-Forward) Phase 2 study
* Have a clinical diagnosis of Tourette Syndrome (TS)
* If using maintenance medication(s) for TS or TS spectrum diagnoses (e.g. obsessive-compulsive disorder [OCD], Attention-Deficit Hyperactivity Disorder [ADHD]), be on stable doses
* Subjects of childbearing potential who do not practice total abstinence must agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently during the screening, treatment and follow-up periods of the study
* Adolescent and adult subjects (12 to 64 years of age) must have a negative urine drug screen for amphetamines, barbiturates, benzodiazepine, phencyclidine, cocaine, opiates, or cannabinoids and a negative alcohol screen. Subjects who are on stable doses of prescribed and supervised (not as needed) benzodiazepines, opiates, or psychostimulants (for subjects with comorbid ADHD) are allowed to participate in the study
* Be in good general health

Exclusion Criteria:

* Have an active, clinically significant unstable medical condition within 1 month prior to screening
* Have a known history of long QT syndrome or cardiac arrhythmia
* Have a known history of neuroleptic malignant syndrome
* Have a cancer diagnosis within 3 years prior to screening (some exceptions allowed)
* Have a blood loss ≥250 mL or donated blood within 56 days prior to screening (subjects 6 to 17 years of age); have a blood loss ≥550 mL or donated blood within 30 days prior to screening (subjects 18 to 64 years of age)
* Have a known history of substance dependence, substance (drug) or alcohol abuse
* Have a significant risk of suicidal or violent behavior
* Have initiated Comprehensive Behavioral Intervention for Tics (CBIT) during the screening period or at baseline or plan to initiate CBIT during the study
* Have received an investigational drug within 30 days before screening or plan to use an investigational drug (other than NBI-98854) during the study

Ages: 6 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 155 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Sun City, Arizona
  - San Diego, California
  - Loxahatchee Groves, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Naperville, Illinois
  - Lincoln, Nebraska
  - Summit, New Jersey
  - New York, New York
  - Norristown, Pennsylvania
  - Nashville, Tennessee
  - Fort Worth, Texas
  - Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled male and female children (6 to 11 years of age), adolescents (12 to 17 years of age), and adults (18 to 64 years of age) from 34 centers in the United States. Participants must have a clinical diagnosis of Tourette Syndrome (TS) and must have previously completed participation in Study NB-98854-1501 or Study NBI-98854-1505. The first and last participant were enrolled on 25 July 2016 and 14 April 2017, respectively.
Period: Overall Study
Arm/Group | Valbenazine (Children) | Valbenazine (Adolescents) | Valbenazine (Adults)
Started | 33 | 41 | 81
Safety Analysis Set (Safety analysis set includes all participants who received at least one dose of study drug and have any postbaseline data.) | 33 | 40 | 79
Completed | 23 | 32 | 49
Not Completed | 10 | 9 | 32
Not completed — Adverse Event | 1 | 2 | 14
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 8 | 6 | 9
Not completed — Lost to Follow-up | 1 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Safety analysis set, which includes all participants who received at least one dose of study drug and have any postbaseline data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Valbenazine (Children) | Valbenazine (Adolescents) | Valbenazine (Adults) | Total
Number analyzed (Participants) | 33 | 40 | 79 | 152
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.5 (1.5) | 13.7 (1.4) | 34.6 (12.9) | 23.6 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 25 | 40
  Male | 26 | 32 | 54 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 4 | 13
  Not Hispanic or Latino | 30 | 34 | 75 | 139
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Asian | 0 | 0 | 1 | 1
  Race: Black or African American | 3 | 2 | 1 | 6
  Race: White | 30 | 35 | 76 | 141
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race: Other | 0 | 1 | 0 | 1
  Race: Multiple | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE is an adverse event not present prior to the initiation of study drug dosing, or is an already present event that worsens either in intensity or frequency following the initiation of study drug dosing.
Time Frame: Baseline through Week 28
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Valbenazine (Children) | Valbenazine (Adolescents) | Valbenazine (Adults)
Number analyzed (Participants) | 33 | 40 | 79
Participants | 20 | 29 | 68

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Arm/Group | Valbenazine (Children) | Valbenazine (Adolescents) | Valbenazine (Adults)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/40 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/40 | 2/79
Other Adverse Events (participants affected / at risk) | 19/33 | 22/40 | 57/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valbenazine (Children) (N=33) | Valbenazine (Adolescents) (N=40) | Valbenazine (Adults) (N=79)
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valbenazine (Children) (N=33) | Valbenazine (Adolescents) (N=40) | Valbenazine (Adults) (N=79)
Nausea (Gastrointestinal disorders) | 2 | 1 | 3
Vomiting (Gastrointestinal disorders) | 3 | 2 | 1
Fatigue (General disorders) | 5 | 4 | 13
Irritability (General disorders) | 4 | 0 | 2
Pyrexia (General disorders) | 2 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 2 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 11
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Protein urine present (Investigations) | 2 | 0 | 0
Weight increased (Investigations) | 2 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Akathisia (Nervous system disorders) | 0 | 1 | 5
Headache (Nervous system disorders) | 5 | 5 | 5
Lethargy (Nervous system disorders) | 2 | 0 | 1
Sedation (Nervous system disorders) | 3 | 8 | 12
Somnolence (Nervous system disorders) | 3 | 8 | 16
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 4
Depression (Psychiatric disorders) | 1 | 0 | 7
Insomnia (Psychiatric disorders) | 2 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI has the right to publish results provided such publication does not violate confidentiality or IP provisions within the contract with the Sponsor. Prior to submission for publication or presentation of results, the PI must provide the Sponsor time for review. The Sponsor can request the PI to withhold or remove information from all publications. For a multi-center study, any publication of results by the PI shall not be made before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT02879578/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT02879578/SAP_001.pdf